CLINICAL TRIAL: NCT03642600
Title: Novel Strategies in Weight Loss in Women With Polycystic Ovary Syndrome: do Changes in the Gut Microbiome Play a Role?
Brief Title: The Gut Microbiome in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S61338
Record Dates: First submitted 2018-08-10; First posted 2018-08-22 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: PCOS; Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — Nutrition Assessment; Inositol; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dietary advice plus myo-inositol and folic acid (Active Comparator): 2gram myo-inositol and folic acid twice daily orally lack of consistent evidence for myo-inositol as treatment of women with PCOS
  Interventions: Dietary Supplement: dietary advice plus myo-inositol and folic acid
- dietary advice plus liraglutide pen injector (Active Comparator): liraglutide starting at 0.6 mg, gradually increasing up to a dose of 3 mg daily after four weeks no evidence for weight loss in women with PCOS
  Interventions: Drug: dietary advice plus Liraglutide Pen Injector

INTERVENTIONS:
Dietary Supplement: dietary advice plus myo-inositol and folic acid — dietary advice and lifestyle interventions and myo-inositol
  Arms: dietary advice plus myo-inositol and folic acid
Drug: dietary advice plus Liraglutide Pen Injector — dietary advice and lifestyle interventions and liraglutide pen injector
  Arms: dietary advice plus liraglutide pen injector

SUMMARY:
Testing two different strategies for weight loss intervention and revealing possible changes in composition of gut microbiota, in order to provide more insight in the effect of dietary changes and weight loss treatments on gut microbiome in overweight and obese women with polycystic ovary syndrome (PCOS). The two strategies are:

* dietary advice plus myo-inositol and folic acid
* dietary advice plus liraglutide, glucagon-like peptide-1 (GLP-1) receptor agonist Primary outcome will be weight loss. Secondary outcomes are longitudinal changes in clinical features associated with PCOS and metabolic syndrome, longitudinal changes in gut microbiome with interventions.

Subjects will be treated during 16 weeks and follow-up will take 16 weeks after stop of treatment.

ELIGIBILITY:
Inclusion Criteria:

* PCOS according to ROtterdam criteria
* BMI ≥ 27 kg/m2 and at risk of metabolic syndrome or BMI ≥ 30 kg/m2

Exclusion Criteria:

* pregnancy
* pancreatitis (in the past)
* oral contraceptive pill use
* inflammatory bowel disease
* auto-immune disease
* immuno-modulatory drugs
* antidiabetic drugs
* anti-inflammatory drugs

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
weight loss | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lie Fong, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- Sharon Lie Fong, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No